CLINICAL TRIAL: NCT06800898
Title: The Methylation Level of the Orexin Gene in Anorexia Nervosa: Relationship With Eating Disorder, Depressive State, and Sleep Quality
Brief Title: Orexin Gene in Anorexia Nervosa
Acronym: ORESSANNE
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 01C414
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Anorexia Nervosa
Keywords: Orexins; Methylation; Epigenetics; Psychiatric comorbidities; Eating disorder; Quality of sleep
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders; Sleep Initiation and Maintenance Disorders | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood sample; with pyrosequencing, the methylation of the promoter of the OX-A and OX-B genes is evaluated using DNA extracted from peripheral nucleated cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anorexia Nervosa: Young women with Anorexia Nervosa, hospitalized at the Division of Eating and Nutrition Disorders, Istituto Auxologico Italiano, IRCCS, Piancavallo, Italy,
  Interventions: Other: Blood samples and Questionnaires
- Normal weight: Young women of comparable age with Body Mass Index between 18.5 and 24.9 kg/m2
  Interventions: Other: Blood samples and Questionnaires

INTERVENTIONS:
Other: Blood samples and Questionnaires — Blood samples for methylation of the promoter of the OX-A and OX-B genes and questionnaires:
  Eating Disorder Examination Q Eating Disorder Inventory 3 Major Depression Inventory Symptom Checklist-revised ESS - Epworth Sleepiness Scale Pittsburgh Sleep Quality Index Horne & Ostberg questionnaire

SUMMARY:
The objectives of this study will be to determine the methylation of the promoter of the Orexin A (OX-A) and B (OX-B) genes in young women (> 18 years) with Anorexia Nervosa (AN), compared with a control group; and to evaluate the relationship of promoter methylation of the genes for OX-A and OX-B with the severity of the eating disorder, psychiatric comorbidities (in particular, depression), and sleep quality.

ELIGIBILITY:
Patients with Anorexia Nervosa:

Inclusion Criteria:

* Female sex
* Age 18 years and older
* Anorexia Nervosa
* Hospitalized at the Division of Eating and Nutrition Disorders, Istituto Auxologico Italiano, IRCCS, Piancavallo, Italy

Exclusion Criteria:

* Absence of signed informed consent

Control group:

Inclusion Criteria:

* Female sex
* Age 18 years and older
* Body Mass Index between 18.5 and 24.9 kg/m2

Exclusion Criteria:

* Absence of signed informed consent
* Presence of any physical and mental pathology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 young women (> 18 years old), hospitalized at the Division of Eating and Nutrition Disorders, Istituto Auxologico Italiano, IRCCS, Piancavallo (VB), for each of whom a diagnosis of AN will be formulated based on the DSM-criteria 5 (Diagnostic and Statistical Manual of Mental Disorders 5; American Psychiatric Association, 2013).
  For each patient, a woman of comparable age, with a BMI between 18.5 and 24.9 kg/m2, is enrolled in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Orexin A promoter methylation | Baseline
  Percentage of Orexin A promoter methylation
Orexin B promoter methylation | Baseline
  Percentage of Orexin B promoter methylation

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Site Piancavallo, Oggebbio, Verbania, Italy